CLINICAL TRIAL: NCT03476148
Title: Effect of Home-Based Rehabilitation Using Interactive Motion Tracking Device on Function and Patient Satisfaction After Total Knee Arthroplasty
Brief Title: Home Rehabilitation Using Interactive Device Versus Inpatient Rehabilitation in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rehab. Home vs inpatient
Record Dates: First submitted 2018-03-13; First posted 2018-03-23 (Actual); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis, Knee; Arthroplasty; Rehabilitation
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive Device Rehabilitation (Experimental)
  Interventions: Device: Home Rehabilitation using Interactive device
- Inpatient Rehabilitation (Active Comparator)
  Interventions: Other: Inpatient Rehabilitation

INTERVENTIONS:
Device: Home Rehabilitation using Interactive device — Rehabilitation is performed using interactive motion tracking augmented reality device. 6 exercises are included in one-day rehabilitation program. Each exercise is recorded in aspect of compliance, completion.
  Arms: Interactive Device Rehabilitation
Other: Inpatient Rehabilitation — Patients are given the exercises in the setting of inpatient rehabilitation
  Arms: Inpatient Rehabilitation

SUMMARY:
Rehabilitation after total knee arthroplasty is very important in terms of range of motion of the knee, muscle power, normal gait, pain control and consequently the patient's satisfaction. Convectional rehabilitation methods in assist of therapist required high demand of resources. Recently, outpatient clinic or tele-communication tool based rehabilitations were investigated and reported equivalent results. However, those methods also required group or one-to-one facing that restricted availability of the exercise.

With development of the motion tracking technology, new device that gives real time feedback with augmented reality images can be used for rehabilitation in home-based setting.

This study aims to compare the clinical outcomes after the rehabilitation by interactive home-based device or conventional inpatient setting.

DETAILED DESCRIPTION:
The objective of this work is to compare the pain, stiffness, function and satisfaction between groups at 6 months after the total knee arthroplasty.

The investigators hypothesized that the clinical outcomes of rehabilitation by interactive home-based device are not inferior than that by conventional inpatient setting.

The study design is a single-blind non-randomized controlled trial. Patients takes different rehabilitation method but the outcome assessor is blinded. The clinical outcome is compared at preoperative, postoperative 6weeks, 3months. And clinical outcome consists of Range of Motion (ROM), WOMAC (Western Ontario and McMaster University Arthritis Index ) score, Knee Society Score, Time-up-go (TUG) test.

ELIGIBILITY:
Inclusion Criteria:

* over 19 year old
* Patients for total knee arthroplasty of one knee
* Patients who can understand and utilize the device

Exclusion Criteria:

* who don't agree with participation of the study
* who can not understand and utilize the device
* Rheumatoid arthritis, Other inflammatory arthritis
* Neuropsychiatric patients

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-22 (Estimated); Primary Completion 2018-12-31 (Estimated); Study Completion 2020-03-21 (Estimated)

PRIMARY OUTCOMES:
Change in Western Ontario and McMaster Universities Index(WOMAC index) | preoperative, postoperative at 6, 12 weeks
Change in Knee Society Score | preoperative, postoperative at 6, 12 weeks
Change in Time-Up-Go (TUG) test | preoperative, postoperative at 6, 12 weeks